CLINICAL TRIAL: NCT02306213
Title: Effect of Hydroxyethylstarch 6% 130/0.4 Administration on Renal Function After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Momeni, MD, PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cliniques Universitaires Saint
Record Dates: First submitted 2014-11-20; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Kidney Function Tests
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

ARMS (2):
- Hydroxyethylstarch 6% 130/0.4 (Experimental): These patients have received Hydroxyethylstarch 6% 130/0.4 intraoperatively or postoperatively in addition to standard volume therapy.
  Interventions: Drug: Hydroxyethylstarch 6% 130/0.4; Other: standard volume therapy
- No Hydroxyethylstarch 6% 130/0.4 (Active Comparator): These patients have not received Hydroxyethylstarch 6% 130/0.4 at any time point. Only standard volume therapy has been used.
  Interventions: Other: standard volume therapy

INTERVENTIONS:
Drug: Hydroxyethylstarch 6% 130/0.4 — Use of Hydroxyethylstarch intraoperatively, for cardiopulmonary bypass use and postoperatively in the intensive care unit
  Other Names: Any volume therapy has been recorded
  Arms: Hydroxyethylstarch 6% 130/0.4
Other: standard volume therapy

SUMMARY:
Recent studies have shown an increased incidence of renal replacement therapy after the use of Hydroxyethylstarchs (HES) in patients admitted in the intensive care unit. However, studies showing detrimental effects of HES have been conducted in mostly non-surgical subjects. There are very few studies analyzing the effects of HES on renal function after cardiac surgery, a population already at risk of renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing cardiac surgery

Exclusion Criteria:

* Heart transplantation
* Ventricular assist devices
* Patients requiring extracorporeal life support before or after cardiac surgery
* Patients revised for bleeding and/or tamponnade presenting with hemodynamic instability
* Patients in whom the administered volume therapy was not completely available
* Subjects who required renal replacement therapy before surgery
* Trauma patients who were put on cardiopulmonary bypass
* Patients who died intra-operatively or soon after arrival in the intensive care unit in whom no postoperative creatinine measurements were available

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1564 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Renal dysfunction based on RIFLE (Risk; Injury; Failure; Loss; End-stage) criteria. | Up to 45 days

SECONDARY OUTCOMES:
Mortality | Up to 45 days